CLINICAL TRIAL: NCT00377429
Title: An Open-Label, Single-Arm, Phase II Safety and Tolerability Study of Catumaxomab (Anti-EpCAM x Anti-CD3) in Women With Advanced Epithelial Ovarian Cancer After a Complete Response to Chemotherapy
Brief Title: Safety and Efficacy Study of Catumaxomab to Treat Ovarian Cancer After a Complete Response to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Collaborators: Fresenius Biotech North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-CAT-OC-01
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Results first posted 2012-07-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Ovarian Cancer
Keywords: Epithelial Cancer; Epithelial Carcinoma; Epithelial Ovarian Cancer; Epithelial Ovarian Carcinoma; Fallopian Tube Cancer; Fallopian Tube Carcinoma; Ovarian Cancer; Ovarian Carcinoma; Ovarian Epithelial Cancer; Ovarian Epithelial Carcinoma; Peritoneal Cancer; Peritoneal Carcinoma; Advanced Epithelial Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- catumaxomab (Experimental)
  Interventions: Drug: catumaxomab

INTERVENTIONS:
Drug: catumaxomab — Catumaxomab administered as four 3-hour, constant-rate, intraperitoneal (IP) infusions of 10, 20, 50, 150 microgram (mcg).
  Other Names: Removab

SUMMARY:
The purpose of this study is to determine whether the investigational drug catumaxomab delivered in the planned treatment schedule is a safe and effective treatment for women with advanced ovarian cancer who experience a complete response to chemotherapy.

DETAILED DESCRIPTION:
A multi-center, phase II study of catumaxomab in ovarian cancer patients who experience a complete response to chemotherapy. Each eligible patient will receive four ascending doses of catumaxomab, administered intraperitoneally via an indwelling catheter or port. Catumaxomab will be administered as a 3-hour constant rate infusion with a dosing interval of 3-4 days. Each patient will participate in this study for up to 4 months (includes the baseline screening period, 11 to 21 days treatment period, and up to 90 days/3 months follow-up), with post-study follow-up every 3 months for 2 years.

Catumaxomab is a trifunctional antibody targeting epithelial cell adhesion molecule (EpCAM) on tumor cells and CD3 (cluster of differentiation 3) on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory cells (e.g. macrophages, dendritic cells [DCs] and natural killer [NK] cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these different immune effector cells, which can trigger a complex anti-tumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form before any protocol-specific screening procedures
* Histologically confirmed diagnosis of epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer, Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) stage IIb - IV
* Optimal or sub-optimal cytoreductive surgery
* Clinical complete response to platinum and taxane-based therapy consisting of at least four cycles, based on computed tomography (CT) scan and a CA-125 (cancer antigen 125) level below 35 U/mL
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Last dose of platinum and taxane-based therapy completed within 6 weeks prior to the start of catumaxomab treatment
* Negative serum pregnancy test result at screening in women of childbearing potential (applies to patients without documented menopause or sterility)
* Willingness of patients of childbearing potential to use an effective contraceptive method (i.e. oral contraceptive, cervical cap, diaphragm with spermicide, condom with spermicide, or intrauterine device) during the study and for at least 6 months after the last infusion

Exclusion Criteria:

* Acute or chronic systemic infection
* Exposure to chemotherapy, radiotherapy, immunotherapy or investigational anti-cancer therapy within 6 weeks of first dose of catumaxomab other than last regimen of platinum and taxane chemotherapy as outlined in protocol
* Known human immunodeficiency virus (HIV) infection
* Previous treatment with non-humanized murine (rat or mouse) monoclonal antibodies (mAb)
* Inadequate renal function (creatinine > 1.5 x upper limit of normal [ULN])
* Inadequate hepatic function:

  * Alanine aminotransferase (ALT) > 2.5 x ULN or
  * Aspartate aminotransferase (AST) > 2.5 x ULN or
  * Bilirubin > 1.5 x ULN
* Platelets < 100,000 cells/mm^3
* Absolute neutrophil count (ANC) < 1,500 cells/mm^3
* History of myocardial infarction, congestive heart failure or relevant cardiac arrhythmia within the last 6 months
* No other malignancy within the past 5 years except non-melanoma skin cancer or carcinoma in situ of the cervix if adequately treated
* No history of brain metastases
* Any further condition or disease that would, in the opinion of the Investigator, expose the patient to undue risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Seiden, MD, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (12):
  - Arizona Cancer Center, Tucson, Arizona
  - Stanford University of Obstetrics and Gynecology, Stanford, California
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Gynecologic Oncology - Hinsdale, Hinsdale, Illinois
  - Michiana Hematology Oncology P.C., South Bend, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Magee-Women Hospital of UPMC, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina

REFERENCES:
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020

RESULTS

PARTICIPANT FLOW:
Groups:
- Catumaxomab: 4 dose series (10-20-50-150 micrograms) within 21 days
Period: Overall Study
Arm/Group | Catumaxomab
Started | 47 (Treated)
Completed | 32 (Completed main study)
Not Completed | 15
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 8
Not completed — Physician Decision | 1
Not completed — Patient non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Catumaxomab
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed a 4-dose Series of Catumaxomab Infusions (Defined as 10-20-50-150 Micrograms) Within 21 Days
Time Frame: 21 days
Population: Treated population
Measure: Number; unit: Participants
Arm/Group | Catumaxomab
Number analyzed (Participants) | 47
Participants | 29

2. Secondary Outcome: Number of Participants With Negative (Undetectable) Humoral Immune Responses to Catumaxomab Therapy
Description: Humoral immune response of participants with functional immune system to catumaxomab can provide important information regarding why a therapy may work for some participants and not for others. An undetectable humoral response by itself does not necessarily imply lack of study drug activity. Humoral response is one of the possible selected measurements of the study drug activity at a time point in the study.
Time Frame: 2 months
Population: Full analysis population
Measure: Number; unit: Participants
Arm/Group | Catumaxomab
Number analyzed (Participants) | 42
Participants | 41

3. Secondary Outcome: Number of Participants With no Residual Disease Prior to Catumaxomab Treatment Via 2nd-look Laparoscopy or Laparotomy (These Procedures Are Optional)
Time Frame: Baseline
Population: 2nd look laparoscopy/laparotomy
Measure: Number; unit: Participants
Arm/Group | Catumaxomab
Number analyzed (Participants) | 11
Participants | 7

4. Secondary Outcome: Median Time of Progression-free Survival in Weeks (Post-study for 24 Months)
Time Frame: 2 years
Population: Post study full analysis set
Measure: Median (Full Range); unit: weeks
Arm/Group | Catumaxomab
Number analyzed (Participants) | 43
weeks | 86.1 [21.3 to 141.0]

5. Secondary Outcome: Number of Participants Who Survived (Post-study at 24 Month Visit)
Description: Number of participants who survived (post-study at 24 month visit) is the number of participants who did not die
Time Frame: 2 years
Population: Post study full analysis set
Measure: Number; unit: participants
Arm/Group | Catumaxomab
Number analyzed (Participants) | 43
participants | 39

6. Secondary Outcome: Number of Participants With no Residual Disease at 3 Months After Catumaxomab Treatment Via 3rd-look Laparoscopy or Laparotomy (These Procedures Are Optional)
Time Frame: 3 months
Population: Only 1 patient received 3rd-look laparoscopy/laparotomy as determined by the investigator and no residual disease was found.
Measure: Number; unit: participants
Arm/Group | Catumaxomab
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Time Frame: End of main study: 90 days after the last dose of study drug
Arm/Group | Catumaxomab
Serious Adverse Events (participants affected / at risk) | 19/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catumaxomab (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Volvulus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Cytokine release syndrome (Immune system disorders) | 5 (5)
Bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes oesophagitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catumaxomab (N=47)
Anaemia (Blood and lymphatic system disorders) | 12 (13)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Tachycardia (Cardiac disorders) | 9 (14)
Nausea (Gastrointestinal disorders) | 38 (79)
Vomiting (Gastrointestinal disorders) | 34 (61)
Abdominal pain (Gastrointestinal disorders) | 33 (59)
Diarrhoea (Gastrointestinal disorders) | 24 (45)
Abdominal distension (Gastrointestinal disorders) | 13 (16)
Constipation (Gastrointestinal disorders) | 10 (13)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5)
Abdominal pain, upper (Gastrointestinal disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 38 (68)
Fatigue (General disorders) | 28 (46)
Chills (General disorders) | 27 (45)
Asthenia (General disorders) | 6 (7)
Pain (General disorders) | 5 (7)
Chest pain (General disorders) | 4 (4)
Malaise (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 4 (4)
Catheter site pain (General disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3)
Cytokine release syndrome (Immune system disorders) | 5 (5)
Urinary tract infection (Infections and infestations) | 8 (8)
Alanine aminotransferase increased (Investigations) | 11 (14)
Blood potassium decreased (Investigations) | 10 (17)
Blood creatinine increased (Investigations) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 7 (8)
Blood alkaline phosphatase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 4 (7)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12)
Anorexia (Metabolism and nutrition disorders) | 9 (10)
Dehydration (Metabolism and nutrition disorders) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 7 (8)
Dizziness (Nervous system disorders) | 5 (6)
Restless legs syndrome (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 15 (19)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Hypotension (Vascular disorders) | 10 (12)
Hypertension (Vascular disorders) | 5 (14)
Flushing (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The 1st publication of study results shall be a multicenter publication or disclosure coordinated by sponsor.

Prior to submitting for publication, the Investigator shall allow sponsor at least 60 days to review the proposed Publication. Proposed Publications shall not include either Fresenius Biotech confidential information other than the study results or personal data on any patient. If parties disagree, parties will meet to discuss and resolve any disagreements.